CLINICAL TRIAL: NCT04895124
Title: Second Follow-up Study of Participants (COPD Patients and Healthy Control Subjects) from the Cross-sectional Study "11-03 Ribolution" for the Evaluation of Predictive Biomarkers Based on Non-coding RNA
Brief Title: Second Follow-up Study of COPD Patients and Healthy Controls for Evaluation of Predictive Non-coding RNA Biomarkers
Acronym: Ribo III
Status: Completed | Type: Observational
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 19-12 Ribolution III
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood, sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Healthy volunteers
- Healthy smokers
- COPD GOLD I
- COPD GOLD II
- COPD GOLD III/IV

SUMMARY:
Between 2012 and 2014, a cohort of 90 COPD subjects of disease severity grades GOLD I-IV as well as 60 healthy control subjects (30 smokers and 30 non-smokers) have been examined regarding different clinical and blood/ sputum derived biomarkers at the investigators' research center.

Of this cohort, 116 subjects were re-invited for the first follow-up study Ribolution II (NTC02522026) after 3 years (+/- 6 months) and data on the clinical course and treatment changes was obtained.

This second follow-up study will re-examine all available subjects regarding disease course and treatment changes after 3 years (+/-6 months) for the investigation of ncRNA/ transcriptome biomarkers for their potential to indicate disease progression. In addition, biobanking of respective biosamples for potential future COPD biomarker research will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in the study "11-03 Ribolution".
2. Able and willing to give written informed consent.
3. Females will be considered for inclusion if they are: not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing.

Exclusion Criteria:

1. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs, lung function or ECG at screening visit, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study.
2. Past or present disease developed after the participation in "11-03 Ribolution" or "15-01 Ribolution II", which might interfere with study procedures.
3. Participation in another clinical trial 30 days prior to enrollment.
4. Current drug or alcohol abuse.
5. Risk of non-compliance with study procedures.
6. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
7. History of an acute infection four weeks prior to the study procedures, including - but not limited to - moderate or severe exacerbation (requiring oral corticosteroid, antibiotics or hospitalization). All courses of oral corticosteroids and antibiotics must be completed at least four weeks prior to all study procedures (with the exception of the informed consent). In case of significant acute infections or moderate or severe exacerbation, the study participation can be split in two separate visits (1. Informed consent visit, 2. Study procedures visit, when subject is fully resolved, at least four weeks after the end of infection/ exacerbation).
8. If performed according to SOP FHI-1-18, positive SARS-CoV-2 rapid antigen test on Day 1. Subjects may be re-screened when confirmatory nucleic acid amplification test was negative or when officially ordered quarantine has ended.
9. Being a vulnerable subject (dependent, in detention or without mental capacity).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic obstructive pulmonary disease (COPD) GOLD stage I to IV, healthy smokers and healthy non-smokers
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Collecting longitudinal patient information by performing a second follow-up visit. | 9 years ± 12 months after completion of the study "11-03 Ribolution"
  Medical history, physical examination, comprehensive lung function and laboratory assessments will be taken and linked respectively with former study data to collate individual clinical courses.
Analysis of exhaled particles | 9 years ± 12 months after completion of the study "11-03 Ribolution"
  Determining airway dimensions by means of time-resolved single breath analysis and collection of exhaled particles for bioanalysis.
Determining predictive power of non-coding RNA patterns | 9 years ± 12 months after completion of the study "11-03 Ribolution"
  Analysis of non-coding RNA from sputum and blood

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Lower Saxony, Germany